CLINICAL TRIAL: NCT01855581
Title: The Incidence and Nature of Adverse Events During Pediatric Sedation for MRI/CT in One Korean University Hospital: Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0923
Record Dates: First submitted 2013-05-09; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Children Requiring Sedation for MRI/CT
MeSH Terms: interventions — Propofol; Ketamine

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- sedation group: Children requiring sedation for MRI/CT
  Interventions: Drug: pediatric sedation (propofol, ketamine, etc)

INTERVENTIONS:
Drug: pediatric sedation (propofol, ketamine, etc) — Presedation assessment was performed by hospitalists and pediatric sedation was performed by protocol in the sedation unit.
  Data on demographics, primary illness, ASA, snoring history, URI symptom, medications used, procedure and recovery times, medication doses, outcomes of anesthesia, airway interventions and adverse events were collected retrospectively.

SUMMARY:
Sedation and anesthesia for diagnostic imaging represents a rapidly growing field of practice, especially in children. Propofol is the most common sedative drug administered for MRI/CT. However, this drug is associated with adverse events, including pulmonary complications, and there has been no report on these complications in Korea.

The investigators reviewed 3739 charts of pediatric patients sedated for MRI/CT between January and November 2012.

In this study, the investigators will report the nature and frequency of adverse events associated with sedation for MRI/CT between January and November 2012.

ELIGIBILITY:
Inclusion Criteria:

* Requiring sedation for MRI/CT, aged 0- 18 years

Exclusion Criteria:

* None

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children requiring sedation for MRI/CT
Sampling Method: Non-Probability Sample
Enrollment: 3739 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 24 hours
  The investigators will review all adverse events that are associated with pediatric sedation for MRI/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Srinivasan M, Turmelle M, Depalma LM, Mao J, Carlson DW. Procedural sedation for diagnostic imaging in children by pediatric hospitalists using propofol: analysis of the nature, frequency, and predictors of adverse events and interventions. J Pediatr. 2012 May;160(5):801-806.e1. doi: 10.1016/j.jpeds.2011.11.003. Epub 2011 Dec 16. PMID 22177990